CLINICAL TRIAL: NCT03325075
Title: A Phase 1, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Immunogenicity of VAL-181388 in Healthy Adults in a Non-endemic Chikungunya Region
Brief Title: Safety, Tolerability, and Immunogenicity of VAL-181388 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAL-181388-P101; W911NF-13-1-0417 (Other Grant/Funding Number: Defense Advanced Research Projects Agency (DARPA))
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Chikungunya Virus
Keywords: VAL-181388; Chikungunya vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAL-181388 (Experimental)
  Interventions: Biological: VAL-181388
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAL-181388 — Escalating dose levels
  Arms: VAL-181388
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety, tolerability, and immunogenicity of VAL-181388 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 49 years of age
* Body mass index between 18 and 35 kilograms (kg)/square meter (m^2)
* In good health as determined by medical history
* Female participants must be non pregnant and non lactating and meet one of the following criteria: a) post menopausal b) surgically sterile, or c) of childbearing potential and agree to use an adequate contraception method
* Male participants must use an acceptable method of birth control through 3 months after the final vaccination
* Agrees to comply with the study procedures and provides written informed consent
* Has access to a consistent and reliable means of telephone contact and agrees to stay in contact with the study site for the duration of the study

Exclusion Criteria:

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* Female of childbearing potential and has a positive pregnancy test at screening or on the day of vaccination
* Abnormal vital signs or screening safety laboratory test results including liver enzyme tests
* Administration of an investigational product within 60 days, or 5 half-lives, whichever is longer
* Administration of any live attenuated vaccines within 4 weeks before enrollment or inactive vaccines within 2 weeks before enrollment, or plans to receive any vaccine during the active vaccination period
* Prior administration of a vaccine for chikungunya virus (CHIKV), dengue, Yellow Fever, tick-borne encephalitis, a history of confirmed or suspected CHIKV infection, or has lived in a CHIKV-endemic area greater than 1 year or cumulative stay of greater than 30 days in 5 years
* Prior administration of investigational agent using formulations similar to VAL-181388
* A history of hypersensitivity or serious reactions to previous vaccinations
* Any known or suspected autoimmune disease or immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination
* A history of inflammatory arthritis
* Any neurologic disorder
* Prior administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study drug or plans to receive such products at any time during the study
* Any chronic administration of an immunosuppressant or other immune modifying drug
* Daily or every other day administration of antipyretic or analgesic medication
* Any acute illness at the time of enrollment
* Any significant disorder of coagulation requiring ongoing or intermittent treatment
* A history of idiopathic urticaria
* A history of alcohol abuse or drug addiction
* A positive test result for drugs of abuse
* The participant has any abnormality or permanent body art (for example, tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study drug or interpretation of study results
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies
* A history of active cancer (malignancy) in the last 10 years
* Donation of blood or blood products >450 milliliters (mL) within 30 days of dosing
* Is an employee or first degree relative of the Sponsor, clinical research organization (CRO), or study site personnel

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optimal Research, Rockville, Maryland, United States

REFERENCES:
- [Derived] Shaw CA, August A, Bart S, Booth PJ, Knightly C, Brasel T, Weaver SC, Zhou H, Panther L. A phase 1, randomized, placebo-controlled, dose-ranging study to evaluate the safety and immunogenicity of an mRNA-based chikungunya virus vaccine in healthy adults. Vaccine. 2023 Jun 13;41(26):3898-3906. doi: 10.1016/j.vaccine.2023.04.064. Epub 2023 May 18. PMID 37210308

RESULTS

PARTICIPANT FLOW:
Groups:
- VAL-181388 Dose A: Participants received 2 intramuscular (IM) injections of VAL-181388 Dose A separated by 28 days.
- VAL-181388 Dose B: Participants received 2 IM injections of VAL-181388 Dose B separated by 28 days.
- VAL-181388 Dose C: Participants received 2 IM injections of VAL-181388 Dose C separated by 28 days.
- Placebo: Participants received 2 IM injections of VAL-181388 matched placebo separated by 28 days.
Period: Part A: Dose Escalation (28 Days)
Arm/Group | VAL-181388 Dose A | VAL-181388 Dose B | VAL-181388 Dose C | Placebo
Started | 15 | 15 | 15 | 15
Received Vaccination 1 | 15 | 15 | 15 | 15
Received Vaccination 2 | 15 | 14 | 14 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Part B: Follow-up (Up to 364 Days)
Arm/Group | VAL-181388 Dose A | VAL-181388 Dose B | VAL-181388 Dose C | Placebo
Started | 15 | 15 | 15 | 15
Completed | 13 | 13 | 15 | 13
Not Completed | 2 | 2 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other than specified | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo).
Groups:
- VAL-181388 Dose A: Participants received 2 IM injections of VAL-181388 Dose A separated by 28 days.
- Total: Total of all reporting groups
Arm/Group | VAL-181388 Dose A | VAL-181388 Dose B | VAL-181388 Dose C | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.45) | 33.0 (6.76) | 32.2 (8.46) | 29.1 (5.18) | 31.6 (7.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 8 | 34
  Male | 8 | 6 | 5 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 1 | 7
  Not Hispanic or Latino | 12 | 13 | 14 | 14 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 7 | 6 | 7 | 6 | 26
  White | 7 | 7 | 7 | 7 | 28
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Any Solicited Adverse Events (AEs) (Local and Systemic Reactogenicity Events)
Description: Solicited AEs, including local and systemic AEs were recorded by participants daily using the memory aid. Solicited local AEs include injection site induration/swelling, injection site tenderness, injection site erythema/redness, and injection site pain. Solicited systemic AEs include body temperature (oral), generalized myalgia (muscle ache or pain), generalized arthralgia (joint ache or pain), headache, fatigue/malaise (unusual tiredness), nausea/vomiting, and diarrhea. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 7 days following each vaccination
Population: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- VAL-181388 Dose A: Vaccination 1: Participants received first IM injection of VAL-181388 Dose A.
- VAL-181388 Dose A: Vaccination 2: Participants received second IM injection of VAL-181388 Dose A.
- VAL-181388 Dose B: Vaccination 1: Participants received first IM injection of VAL-181388 Dose B.
- VAL-181388 Dose B: Vaccination 2: Participants received second IM injection of VAL-181388 Dose B.
- VAL-181388 Dose C: Vaccination 1: Participants received first IM injection of VAL-181388 Dose C.
- VAL-181388 Dose C: Vaccination 2: Participants received second IM injection of VAL-181388 Dose C.
- Placebo: Vaccination 1: Participants received first IM injection of VAL-181388 matched placebo.
- Placebo: Vaccination 2: Participants received second IM injection of VAL-181388 matched placebo.
Arm/Group | VAL-181388 Dose A: Vaccination 1 | VAL-181388 Dose A: Vaccination 2 | VAL-181388 Dose B: Vaccination 1 | VAL-181388 Dose B: Vaccination 2 | VAL-181388 Dose C: Vaccination 1 | VAL-181388 Dose C: Vaccination 2 | Placebo: Vaccination 1 | Placebo: Vaccination 2
Number analyzed (Participants) | 15 | 15 | 14 | 13 | 15 | 14 | 15 | 15
Participants | 11 | 10 | 11 | 10 | 13 | 12 | 7 | 5

2. Primary Outcome: Part A: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent AE (TEAE) was defined as any event not present before exposure to vaccine or any event already present that worsens in intensity or frequency after exposure. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 28 days following each vaccination
Population: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | VAL-181388 Dose A: Vaccination 1 | VAL-181388 Dose A: Vaccination 2 | VAL-181388 Dose B: Vaccination 1 | VAL-181388 Dose B: Vaccination 2 | VAL-181388 Dose C: Vaccination 1 | VAL-181388 Dose C: Vaccination 2 | Placebo: Vaccination 1 | Placebo: Vaccination 2
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 15
Participants | 4 | 3 | 6 | 3 | 3 | 6 | 8 | 6

3. Primary Outcome: Part A: Number of Participants With Serious AEs (SAEs), Medically-Attended AEs, and AEs of Special Interest
Description: An MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner (HCP). An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AEs of special interest were evaluated as defined in the protocol. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 28 days following each vaccination
Population: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | VAL-181388 Dose A: Vaccination 1 | VAL-181388 Dose A: Vaccination 2 | VAL-181388 Dose B: Vaccination 1 | VAL-181388 Dose B: Vaccination 2 | VAL-181388 Dose C: Vaccination 1 | VAL-181388 Dose C: Vaccination 2 | Placebo: Vaccination 1 | Placebo: Vaccination 2
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 15
Participants
  SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Medically-Attended AEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AEs of Special Interest | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With SAEs and AEs of Special Interest
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AEs of special interest were evaluated as defined in the protocol. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Through 1 year following the last vaccination
Population: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- VAL-181388 Dose A: Participants who received VAL-181388 Dose A in Part A, were followed up for longer-term safety and immune persistence in Part B.
- VAL-181388 Dose B: Participants who received VAL-181388 Dose B in Part A, were followed up for longer-term safety and immune persistence in Part B.
- VAL-181388 Dose C: Participants who received VAL-181388 Dose C in Part A, were followed up for longer-term safety and immune persistence in Part B.
- Placebo: Participants who received VAL-181388 matched placebo in Part A, were followed up for longer-term safety and immune persistence in Part B.
Arm/Group | VAL-181388 Dose A | VAL-181388 Dose B | VAL-181388 Dose C | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  SAEs | 0 | 0 | 1 | 0
  AEs of Special Interest | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through 1 year following the last vaccination
Description: The safety analysis set included all participants who received at least 1 dose of study drug (VAL-181388 or placebo).
Groups:
- Part A - VAL-181388 Dose A: Vaccination 1: Participants received first IM injection of VAL-181388 Dose A.
- Part A - VAL-181388 Dose A: Vaccination 2: Participants received second IM injection of VAL-181388 Dose A.
- Part A - VAL-181388 Dose B: Vaccination 1: Participants received first IM injection of VAL-181388 Dose B.
- Part A - VAL-181388 Dose B: Vaccination 2: Participants received second IM injection of VAL-181388 Dose B.
- Part A - VAL-181388 Dose C: Vaccination 1: Participants received first IM injection of VAL-181388 Dose C.
- Part A - VAL-181388 Dose C: Vaccination 2: Participants received second IM injection of VAL-181388 Dose C.
- Part A - Placebo: Vaccination 1: Participants received first IM injection of VAL-181388 matched placebo.
- Part A - Placebo: Vaccination 2: Participants received second IM injection of VAL-181388 matched placebo.
- Part B - VAL-181388 Dose A: Participants who received VAL-181388 Dose A in Part A, were followed up for longer-term safety and immune persistence in Part B.
- Part B - VAL-181388 Dose B: Participants who received VAL-181388 Dose B in Part A, were followed up for longer-term safety and immune persistence in Part B.
- Part B - VAL-181388 Dose C: Participants who received VAL-181388 Dose C in Part A, were followed up for longer-term safety and immune persistence in Part B.
- Part B - Placebo: Participants who received VAL-181388 matched placebo in Part A, were followed up for longer-term safety and immune persistence in Part B.
Arm/Group | Part A - VAL-181388 Dose A: Vaccination 1 | Part A - VAL-181388 Dose A: Vaccination 2 | Part A - VAL-181388 Dose B: Vaccination 1 | Part A - VAL-181388 Dose B: Vaccination 2 | Part A - VAL-181388 Dose C: Vaccination 1 | Part A - VAL-181388 Dose C: Vaccination 2 | Part A - Placebo: Vaccination 1 | Part A - Placebo: Vaccination 2 | Part B - VAL-181388 Dose A | Part B - VAL-181388 Dose B | Part B - VAL-181388 Dose C | Part B - Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 0/14 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 1/14 | 0/15 | 0/15 | 0/15 | 0/15 | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 3/15 | 6/15 | 3/14 | 3/15 | 6/14 | 8/15 | 6/15 | 0/15 | 0/15 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - VAL-181388 Dose A: Vaccination 1 (N=15) | Part A - VAL-181388 Dose A: Vaccination 2 (N=15) | Part A - VAL-181388 Dose B: Vaccination 1 (N=15) | Part A - VAL-181388 Dose B: Vaccination 2 (N=14) | Part A - VAL-181388 Dose C: Vaccination 1 (N=15) | Part A - VAL-181388 Dose C: Vaccination 2 (N=14) | Part A - Placebo: Vaccination 1 (N=15) | Part A - Placebo: Vaccination 2 (N=15) | Part B - VAL-181388 Dose A (N=15) | Part B - VAL-181388 Dose B (N=15) | Part B - VAL-181388 Dose C (N=15) | Part B - Placebo (N=15)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - VAL-181388 Dose A: Vaccination 1 (N=15) | Part A - VAL-181388 Dose A: Vaccination 2 (N=15) | Part A - VAL-181388 Dose B: Vaccination 1 (N=15) | Part A - VAL-181388 Dose B: Vaccination 2 (N=14) | Part A - VAL-181388 Dose C: Vaccination 1 (N=15) | Part A - VAL-181388 Dose C: Vaccination 2 (N=14) | Part A - Placebo: Vaccination 1 (N=15) | Part A - Placebo: Vaccination 2 (N=15) | Part B - VAL-181388 Dose A (N=15) | Part B - VAL-181388 Dose B (N=15) | Part B - VAL-181388 Dose C (N=15) | Part B - Placebo (N=15)
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03325075/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT03325075/SAP_001.pdf
  • Informed Consent Form (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03325075/ICF_002.pdf